CLINICAL TRIAL: NCT03837067
Title: Use and Misuse of Domperidone in Parkinson's Disease in France - Dump Investigation
Acronym: DUMP-invest
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: DUMP
Record Dates: First submitted 2018-12-12; First posted 2019-02-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2018-07

CONDITIONS: Parkinson's Disease
Keywords: Domperidone
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson disease is the second most frequent neurodegenerative disease after Alzheimer disease and affect 1% of the population over 60 years. The treatment of PD is based on dopamine replacement therapies (DRT). Nausea is the most frequent adverse event whatever the drug, occurring in 30-40% of patients at the initiation of DRT.

Domperidone, a dopamine D2 receptor antagonist with antiemetic properties, does not readily cross the blood-brain barrier, allowing its used in PD. Domperidone may prolong the duration of the QT interval in predisposed patients, and has been associated with proarrhythmia and arrhythmic deaths. Arrhythmias, sudden death and cardiac arrest were reported with high intravenous doses which has led to withdraw of the parenteral form of the drug in 1984. Two case control studies found an increased risk of sudden death associated with domperidone use. In these reports, the increased risk was depending on age, dose, and the use of domperidone in combination with CYP3A4 inhibitors. Following the discussion created by this alert, the PRAC of the EMA has issued recommendations restricting domperidone use to patients younger than 60 years at doses below 30 mg/day and for a short period (7 days).

Because there is no alternative antiemetic drug to be used in PD, domperidone is commonly prescribed as a preventive therapy in most PD patients initiating DRT. In this population, usually older than 60 years, doses of 60 or 80 mg/day are commonly prescribed, for at least 2 months of the DRT escalating dose period or longer. A particular "niche" of domperidone misuse might be patients treated with continuous subcutaneous administration of apomorphine, a second line therapy in PD, inducing severe and prolonged nausea in almost all patients. Little is known about the use of domperidone in PD in France, but misuse of domperidone in PD patients is probably very high. Data collected from two French PD cohorts, COPARK and DIGPD, showed that 8-14% of PD patients were treated with domperidone.

The aim of this proposal is to investigate the practices and beliefs of French neurologists regarding use and misuse of domperidone in PD, by a qualitative approach.

DETAILED DESCRIPTION:
Parkinson disease is the second most frequent neurodegenerative disease after Alzheimer disease and affect 1% of the population over 60 years (150 to 170 000 patients in France). The treatment of PD is based on dopamine replacement therapies (DRT). Nausea is the most frequent adverse event whatever the drug, occurring in 30-40% of patients at the initiation of DRT.

Domperidone is a dopamine D2 receptor antagonist with antiemetic properties. Domperidone does not readily cross the blood-brain barrier, allowing its used in PD. Domperidone may prolong the duration of the QT interval in predisposed patients, and has been associated with proarrhythmia and arrhythmic deaths. Arrhythmias, sudden death and cardiac arrest were reported with high intravenous doses which has led to withdraw of the parenteral form of the drug in 1984. More recently, two case control studies found an increased risk of sudden death associated with domperidone use. In these reports, the increased risk was depending on age, dose, and the use of domperidone in combination with CYP3A4 inhibitors. Following the discussion created by this alert, the Pharmacovigilance Risk Assessment Committee (PRAC) of the European Medicines Agency (EMA) has issued recommendations restricting domperidone use to patients younger than 60 years at doses below 30 mg/day and for a short period (7 days).

Because there is no alternative antiemetic drug to be used in PD, domperidone is commonly prescribed as a preventive therapy in most PD patients initiating DRT since more than 30 years. In this population, usually older than 60 years, doses of 60 or 80 mg/day are commonly prescribed, for at least 2 months of the DRT escalating dose period or longer. A particular "niche" of domperidone misuse might be patients treated with continuous subcutaneous administration of apomorphine, a second line therapy in PD, inducing severe and prolonged nausea in almost all patients. Little is known about the use of domperidone in PD in France in clinical practice, but misuse of domperidone in PD patients is probably very high. Data collected from two French PD cohorts, COPARK and DIGPD, showed that 8-14% of PD patients were treated with domperidone, extrapolating 10,000 to 20,000 potentially exposed patients at particularly high risk of sudden death.

The aim of this proposal is to investigate the practices and beliefs of French neurologists regarding use and misuse of domperidone in PD, by a qualitative approach. Practices of domperidone prescription by neurologists (from university and general hospitals and private offices) will be evaluated using a semi-structured questionnaire survey. This qualitative study will provide insights from the neurologists on their need for domperidone, therapeutic alternatives and their perceived efficacy, and on the domperidone management and safety procedures that are applied to PD patients before and after domperidone prescription.

The results of this survey on regular practices of neurologists on the use and misuse of domperidone will provide information of the current opinions about the drug, the indications for which it is prescribed, how contra-indications are evaluated, and their feedback on tolerance and efficacy. This information will help Regulatory Authorities to communicate about the safety profile of the drug.

ELIGIBILITY:
Inclusion Criteria:

* All neurologists in France

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All neurologists in France
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Practices of domperidone prescription by neurologists | day 1
  Practices of domperidone prescription by neurologists : use and misuse of domperidone evaluated using a semi-structured questionnaire survey

CONTACTS AND LOCATIONS:
Locations (1):
- La Pitié Salpétrière Hospital, Paris, France